CLINICAL TRIAL: NCT00149799
Title: Pharmacotherapy Relapse Prevention in Body Dysmorphic Disorder
Brief Title: Effectiveness of Escitalopram in the Treatment of Body Dysmorphic Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH072854 (NIH); R01MH072854 (NIH); 2004-P-002305 (Other: IRB Protocol Number); DSIR 83-ATSO
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Anxiety Disorders; Somatoform Disorders
Keywords: Body Dysmorphic Disorder; Escitalopram; Lexapro; BDD; Body Image
MeSH Terms: conditions — Anxiety Disorders; Somatoform Disorders; Body Dysmorphic Disorders | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Experimental): In Phase I, all participants received open-label escitalopram for 14 weeks (at a dosage of 10 mg/d in weeks 1-3, 20 mg/d weeks 4-6, and 30 mg/d thereafter). Participants who responded to escitalopram in Phase I of the study (Weeks 1-14) were randomized to continue with escitalopram for Phase II of the study (Weeks 16-40)
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Participants who responded to escitalopram in Phase I of the study (Weeks 1-14) were randomized to receive a placebo for Phase II of the study (Weeks 16-40)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — At the end of the initial 14-week phase (open-label escitalopram), participants who responded to open-label escitalopram were randomly assigned to receive escitalopram (same dose as received in Phase I) for an additional 6 months.
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Placebo — At the end of the initial 14-week phase (open-label escitalopram), participants who responded to open-label escitalopram were randomly assigned to receive placebo for an additional 6 months.
  Arms: Placebo

SUMMARY:
This study's primary aim is to compare time to relapse and relapse rates in responders to acute escitalopram who are then randomized to placebo versus continuation treatment with escitalopram.

DETAILED DESCRIPTION:
We propose to conduct the first pharmacotherapy relapse prevention study in body dysmorphic disorder (BDD). BDD, an often-delusional preoccupation with a nonexistent or slight defect in appearance, is a distressing, impairing, and common body image disorder. It is associated with high rates of functional impairment and markedly poor quality of life. It appears that serotonin reuptake inhibitors (SRIs) are often--and selectively--efficacious for BDD and that many BDD patients receive SRIs. It also appears that most patients discontinue an efficacious SRI at some point, as the alternative is life-long treatment. However, no relapse prevention studies have been done. Such a study is important from a clinical and public health perspective, because BDD appears to often be chronic and require long-term treatment. It is therefore critically important to investigate the risk of relapse with SRI discontinuation, and whether continuation SRI treatment decreases relapse risk.

Subjects will be enrolled and first treated openly for 14 weeks with escitalopram; 58 escitalopram responders will then be randomized to double-blind continuation treatment with escitalopram or placebo for 6 additional months. Our primary aim is to compare time to relapse and relapse rates in responders to acute escitalopram who are then randomized to placebo versus continuation treatment with escitalopram. Secondary/exploratory aims will explore 1) Whether subjects who receive continuation escitalopram perform better on secondary outcome measures (e.g., quality of life) than those on placebo; 2) Change in symptoms with continuation of escitalopram during the continuation phase; and 3) Acute treatment response.

In summary, this study will be the first relapse prevention study in BDD and the first study of continuation pharmacotherapy in BDD. It will provide critically important information on relapse with continuation versus discontinuation of an SRI, whether continuation treatment protects against relapse, and change in symptoms with continuation treatment. This study will yield unique and clinically important data, and will fill gaps in knowledge about this common, severe, and understudied illness.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient men and women age 18 and older
* Diagnosis of BDD within 6 months of study start date based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)
* Score of 24 or higher on the BDD-Yale-Brown Obsessive Compulsive Scale
* Lives within driving distance of Boston, MA or Providence, RI

Exclusion Criteria:

* Suicidal or homicidal tendencies
* Alcohol/drug abuse or dependence within 3 months of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, PhD, Principal Investigator — Massachusetts General Hospital (MGH); Katharine Phillips, MD, Principal Investigator — Rhode Island Hospital (RIH)
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Fang A, Porth R, Phillips KA, Wilhelm S. Personality as a Predictor of Treatment Response to Escitalopram in Adults With Body Dysmorphic Disorder. J Psychiatr Pract. 2019 Sep;25(5):347-357. doi: 10.1097/PRA.0000000000000415. PMID 31505519
- [Derived] Weingarden H, Shaw AM, Phillips KA, Wilhelm S. Shame and Defectiveness Beliefs in Treatment Seeking Patients With Body Dysmorphic Disorder. J Nerv Ment Dis. 2018 Jun;206(6):417-422. doi: 10.1097/NMD.0000000000000808. PMID 29557815
- See also: Click here to go to the official website of the Body Dysmorphic Disorder Clinic at MGH — http://www.mghocd.org/bdd

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 100 participants received open-label escitalopram in Phase I. Only those who completed Phase I, met criteria for response, and were willing to continue on in the study were subsequently randomized in Phase II (n=58).
Groups:
- Phase I: Open-Label Escitalopram: Participants taking 14 weeks of open-label escitalopram. Subjects received 10 mg/d weeks 1-3, 20 mg/d weeks 4-6, and 30 mg/d thereafter.
- Phase II: Double-blind Escitalopram: At the end of the initial 14-week phase, participants who responded to open-label escitalopram were randomly assigned to receive escitalopram (same dose as received in Phase I) for an additional 6 months.
- Phase II: Double-blind Placebo: At the end of the initial 14-week phase, participants who responded to open-label escitalopram were randomly assigned to receive placebo for an additional 6 months.
Period: Open Label Escitalopram (Phase I)
Arm/Group | Phase I: Open-Label Escitalopram | Phase II: Double-blind Escitalopram | Phase II: Double-blind Placebo
Started | 100 | 0 | 0
Completed | 74 (14 completers were non-responders and 2 responders terminated the study after completing Phase I) | 0 | 0
Not Completed | 26 | 0 | 0
Period: Discontinuation (Phase II)
Arm/Group | Phase I: Open-Label Escitalopram | Phase II: Double-blind Escitalopram | Phase II: Double-blind Placebo
Started | 0 | 28 (Only responders who completed Phase I and were willing to continue were randomized in Phase II) | 30 (Only responders who completed Phase I and were willing to continue were randomized in Phase II)
Completed | 0 | 25 | 21
Not Completed | 0 | 3 | 9

BASELINE CHARACTERISTICS:
Population: As the primary endpoint is based on participants randomized to Phase II (i.e. those who completed Phase I, met criteria for response, and were willing to continue on in the study), baseline characteristics are provided for the 58 Phase II participants.
Groups:
- Phase II: Escitalopram: At the end of the initial 14-week phase, participants who responded to open-label escitalopram were randomly assigned to receive escitalopram (same dose as received in Phase I) for an additional 6 months.
- Phase II: Placebo: At the end of the initial 14-week phase, participants who responded to open-label escitalopram were randomly assigned to receive placebo for an additional 6 months.
- Total: Total of all reporting groups
Arm/Group | Phase II: Escitalopram | Phase II: Placebo | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (12.4) | 31.8 (13.5) | 33.5 (12.4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 27 | 28 | 55
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 24 | 27 | 51
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 58

OUTCOME MEASURES:

1. Primary Outcome: Phase II Relapse of Body Dysmorphic Disorder (BDD) Symptoms (as Measured by the BDD-YBOCS)
Description: We compared the rate of relapse (accounting for time from randomization to relapse and censoring) by treatment arm in Phase II.
Time Frame: Phase II: Biweekly for six months after randomization
Population: Intent-to-treat analysis of all 58 patients randomized to Phase II.
Measure: Number; unit: percentage of subjects who relapsed
Arm/Group | Phase II: Escitalopram | Phase II: Placebo
Number analyzed (Participants) | 28 | 30
percentage of subjects who relapsed | 18 | 40
Statistical Analysis 1: Comparison: Phase II: Escitalopram vs Phase II: Placebo; Cox proportional hazards regression was used to compare relapse rates (accounting for censoring and time from randomization to relapse) in Phase II; Test type: Superiority or Other; p = 0.048, Regression, Cox; p-value is based on the likelihood ratio Chi-Square statistic; Hazard Ratio (HR) = 2.73, 95% CI 2-sided [1.01 to 8.59]

2. Secondary Outcome: Phase I Response to Escitalopram (as Measured by the BDD-YBOCS)
Description: We calculated the proportion of patients who achieved response in Phase I, defined as a >=30% reduction in BDD-YBOCS total score from baseline through the last phase 1 visit.
Time Frame: Phase I: Weekly for weeks 1-4, biweekly from weeks 6-14
Measure: Number; unit: percentage of subjects who responded
Arm/Group | Phase I: Open-Label Escitalopram
Number analyzed (Participants) | 100
percentage of subjects who responded | 67

3. Secondary Outcome: Change in Depression Symptoms (HAM-D) During the Double-blind Relapse Prevention Phase of the Trial (Phase II)
Description: Depressive symptoms were assessed with the Hamilton Rating Scale for Depression (HAM-D), a widely used 21-item depression scale. Of the 21 items on the scale, only the first 17 are used to calculate the total score. Eight of these items are scored on a 5-point scale, ranging from 0 (not present) to 4 (severe symptom), and nine are scored from 0-2. The total score ranges from 0 to 50, where higher scores indicate a greater severity of depression and scores greater than 19 are generally considered indicative of severe depression.
Time Frame: Measured bi-weekly in phase 2 from week 14 (start of randomization for relapse prevention) to week 40
Population: A total of 58 participants who had responded to open-label Escitalopram (phase 1) were randomized to receive either Escitalopram (n=28) or placebo (n=30) in the double-blind relapse prevent trial (phase 2). Some of the assessments visits were missed due to patient cancellations or study dropouts. The exact numbers analyzed are as specified below.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase II: Escitalopram | Phase II: Placebo
Number analyzed (Participants) | 28 | 30
units on a scale
  Week 14: number analyzed (Participants) | 28 | 29
  Week 14 | 3.5357143 (4.4010280) | 3.3793103 (3.3744184)
  Week 16 | 3.8928571 (4.1840906) | 4.2333333 (3.9799786)
  Week 18: number analyzed (Participants) | 28 | 27
  Week 18 | 5.2857143 (5.5099717) | 6.3703704 (6.4875511)
  Week 20: number analyzed (Participants) | 26 | 28
  Week 20 | 4.8461538 (5.5403416) | 5.4285714 (4.7798076)
  Week 22: number analyzed (Participants) | 26 | 27
  Week 22 | 4.2307692 (3.5922995) | 3.7407407 (3.0457106)
  Week 24: number analyzed (Participants) | 25 | 23
  Week 24 | 3.625 (3.3337862) | 3.7727273 (3.0539875)
  Week 26: number analyzed (Participants) | 24 | 25
  Week 26 | 3.8695652 (4.0486176) | 4.04 (3.8457769)
  Week 28: number analyzed (Participants) | 25 | 23
  Week 28 | 4.48 (5.0259327) | 4.4090909 (3.4731499)
  Week 30: number analyzed (Participants) | 23 | 23
  Week 30 | 2.85 (3.9373381) | 4.5454545 (4.0676104)
  Week 32: number analyzed (Participants) | 23 | 22
  Week 32 | 2.9565217 (3.067102) | 4.2 (4.007887)
  Week 34: number analyzed (Participants) | 25 | 21
  Week 34 | 3.375 (3.2412088) | 4.7 (4.5664682)
  Week 36: number analyzed (Participants) | 25 | 22
  Week 36 | 4.0416667 (3.9943348) | 5.4 (5.2555735)
  Week 38: number analyzed (Participants) | 23 | 15
  Week 38 | 3.8181818 (3.8623502) | 3.4666667 (3.8705235)
  Week 40: number analyzed (Participants) | 25 | 19
  Week 40 | 4.2400000 (4.8500859) | 4.1578947 (5.0250833)
Statistical Analysis 1: Comparison: Phase II: Escitalopram vs Phase II: Placebo; We compared change in depression over time by randomized treatment group (Escitalopram vs. Placebo) using a random coefficient model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of change in depression symptom severity in the Escitalopram group will not be significantly different from the placebo group [to be tested]; Test type: Superiority; p = 0.0930, Mixed Models Analysis — A priori threshold for statistical significance: 0.0167 Model term of interest: treatment by time interaction (i.e., slope difference between treatments over time); Degrees of freedom=556; Slope difference = -0.07006, Standard Error of Mean 0.04163

4. Secondary Outcome: Change in Functional Impairment Symptoms (LIFE-RIFT) Over Double-blind Relapse Prevention Phase of the Trial (Phase II)
Description: Subjects switched to placebo were compared to those remaining on escitalopram (double-blind randomization) to assess functional impairment as measured by the Longitudinal Interval Followup Evaluation - Range of Impaired Functioning Tool (LIFE-RIFT). The tool assesses psychosocial functioning in multiple domains, consisting of 5- to 7-point clinician administered scales that obtain information about work, household duties, student work, relationships with family and friends, recreation, life satisfaction, and global social adjustment. Scores can range from 3-22 with higher scores indicating poorer functioning.
Time Frame: Measured three times throughout phase 2 of study (Weeks 14, 28 and 40)
Population: 28 in Escitalopram and 30 were randomized to Placebo after phase-1 open label. Some of the assessments visits were missed due to patient cancellations or study dropouts. The exact numbers analyzed are as specified below. Note: each participant included (28 Escitalopram, 30 placebo) was assessed at least once during phase 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase II: Escitalopram | Phase II: Placebo
Number analyzed (Participants) | 28 | 30
units on a scale
  Week 14: number analyzed (Participants) | 28 | 29
  Week 14 | 9.0000000 (2.6943013) | 8.2413793 (2.3551641)
  Week 28: number analyzed (Participants) | 25 | 23
  Week 28 | 9.8000000 (3.3040379) | 9.0000000 (2.7961012)
  Week 40: number analyzed (Participants) | 25 | 19
  Week 40 | 9.7600000 (3.6887215) | 8.8947368 (3.1428002)
Statistical Analysis 1: Comparison: Phase II: Escitalopram vs Phase II: Placebo; We compared change in functional impairment over time during trial phase 2 by treatment group (Escitalopram vs. Placebo) using a random coefficient model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of change in functional impairment in the Escitalopram group will not be significantly different from that of the placebo group [to be tested]; Test type: Superiority; p = 0.9766, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Degrees of freedom=43; Slope difference = 0.001176, Standard Error of Mean 0.03991

5. Secondary Outcome: Change in Quality of Life (Q-LES-Q-SF) Over Double-blind Relapse Prevention Phase of the Trial (Phase II)
Description: Subjects switched to placebo were compared to those remaining on escitalopram (double-blinded randomization) to assess quality of life changes as measured by the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF). The Q-LES-Q-SF is designed to help assess the degree of enjoyment and satisfaction experienced during the past week across several domains: social, leisure, household, work, emotional well-being, physical, and school; it consists of 5-point rater-administered questions. Raw scores can range from 14-70, which are converted to percentage maximum possible by calculating: % Max = (Raw-minimum score)/(maximum score-minimum score). Q-LES_Q-SF percent scores can range from 0-100, with higher scores indicating greater quality of life and satisfaction.
Time Frame: Measured three times throughout phase 2 of study (Weeks 14, 28 and 40)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage score
Arm/Group | Phase II: Escitalopram | Phase II: Placebo
Number analyzed (Participants) | 28 | 30
Percentage score
  Week 14: number analyzed (Participants) | 28 | 27
  Week 14 | 74.1785714 (12.9930282) | 70.9259259 (16.0166402)
  Week 28: number analyzed (Participants) | 22 | 19
  Week 28 | 70.2727273 (14.1528453) | 67.3684211 (16.0665648)
  Week 40: number analyzed (Participants) | 24 | 17
  Week 40 | 69.0833333 (18.5376624) | 68.6470588 (15.2436100)
Statistical Analysis 1: Comparison: Phase II: Escitalopram vs Phase II: Placebo; We compared change in Q-LES-Q-SF percent scores over time by randomized treatment group (Escitalopram vs. Placebo) using a random coefficient model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of change in Q-LES-Q-SF percent scores in the Escitalopram group will not be significantly different from that of the placebo group [to be tested]; Test type: Superiority; p = 0.7724, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Degrees of freedom=36; Slope difference = 0.05723, Standard Error of Mean 0.1963

ADVERSE EVENTS:
Time Frame: Phase I: Weekly for weeks 1-4, biweekly from weeks 6-14; Phase II: Biweekly for six months after randomization
Arm/Group | Phase I: Open-Label Escitalopram | Phase II: Escitalopram | Phase II: Placebo
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 89/100 | 22/28 | 21/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Open-Label Escitalopram (N=100) | Phase II: Escitalopram (N=28) | Phase II: Placebo (N=30)
Fatigue (General disorders) | 42 (55) | 6 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 36 (43) | 3 (4) | 4 (4)
Sexual Dysfunction (Reproductive system and breast disorders) | 31 (33) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 34 (37) | 3 (4) | 7 (7)
Dry Mouth (General disorders) | 28 (30) | 1 (1) | 3 (3)
Headache (General disorders) | 41 (58) | 9 (18) | 9 (16)
Change in Appetite (Metabolism and nutrition disorders) | 23 (25) | 1 (1) | 3 (3)
Agitation (Psychiatric disorders) | 12 (13) | 0 (0) | 1 (2)
Dizziness (General disorders) | 6 (6) | 1 (1) | 6 (6)
Irritability (Psychiatric disorders) | 6 (6) | 2 (2) | 4 (4)
Sweating (General disorders) | 8 (11) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 10 (10) | 2 (4) | 1 (1)
Somnolence (Psychiatric disorders) | 8 (9) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (11) | 5 (9) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 7 (7) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (9) | 1 (1) | 2 (2)
Cold Symptoms (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 4 (6) | 3 (4)
Indigestion (Gastrointestinal disorders) | 4 (5) | 2 (2) | 0 (0)
Vivid Dreams (General disorders) | 5 (5) | 2 (2) | 0 (0)
Menstrual Cramps (Reproductive system and breast disorders) | 3 (4) | 2 (2) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
Hot Flashes (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Yawning (General disorders) | 5 (5) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Heart Palpitations (Cardiac disorders) | 2 (2) | 1 (2) | 2 (2)
Poison Ivy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Restless Sleep / Not Insomnia (General disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Our findings may not be fully generalizable - for example, we excluded those with a co-occurring substance use disorder, higher levels of suicidality, and more severely ill patients who required concomitant therapy or a higher level of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No